CLINICAL TRIAL: NCT03400553
Title: Time Gain of Pre-hospital Troponin Point of Care Testing in the Diagnosis of an Acute Myocardial Infarction
Brief Title: Troponin POCT in the Diagnosis of an Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Dieter Mesotten, MD, Ziekenhuis Oost-Limburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Troponin-T POCT
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Acute Myocardial Infarction; Troponin
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- non-traumatic thoracic pain (Experimental): Patients with out-of-hospital non-traumatic thoracic pain admitted to the emergency unit via ambulance or MUG will be screened for enrolment. Blood analysis for troponin-T will be performed by 3 different devices as explained earlier.
  Interventions: Diagnostic Test: Blood analysis

INTERVENTIONS:
Diagnostic Test: Blood analysis — The blood of the patients will be analyzed for troponin T measured with 3 different devices: 1) a point-of-care (POC) test performed in the ambulance or MUG, a handheld cobas h232 POC system® (Roche Diagnostics, Switzerland), 2) a POC test at the emergency room, a table top AQT90 FLEX® (Radiometer, The Netherlands) and 3) a central laboratory test performed on cobas® 8000 (Roche Diagnostics, Switzerland).

SUMMARY:
Thoracic pain can be caused by a life threatening disease as for instance a heart attack. Fast diagnosis and treatment is necessary for an advantageous clinical outcome. When a patient enters the emergency unit, an electrocardiogram (ECG) can diagnose a heart attack by recording the electrical activity of the patients' heart. However, an increasing number of patients with an acute myocardial infarction (AMI) are presenting without significant abnormalities on ECG In the latter group, diagnosis is dependent of elevated biochemical markers of myocardiocyte necrosis in the blood such as troponin. Generally, troponins are determined in blood and are analyzed by radiometry or at the hospital's laboratory. Time loss in the acquisition of troponin levels can occur during the workflow due to blood sampling difficulties, transport of the blood samples, processing in the laboratory, and processes inherent to the measuring assays. Roche developed a portable point-of-care (POC) device that determines troponin-T in a few minutes by using small volumes of the patient's blood with the added value that this device can be used in a pre-hospital setting which might save a significant amount of time in determining troponin levels.In this way, a faster diagnosis of AMI can be made improving patients' outcome.

DETAILED DESCRIPTION:
In this prospective pilot study, 70 patients will be recruited over a time period of one year, with non-traumatic thoracic pain in a pre-hospital setting. While the ambulance or MUG is transporting such a patient, he/she is asked (informed consent) if an extra blood sample can be taken for measuring troponin levels by the portable device of Roche (cobas h232®). This can be done during the same venipuncture needed for standard-of-care analysis of the two other blood samples used for troponin-T by the radiometer and the laboratory. An ECG is performed in the ambulance and when it is positive, a patient is diagnosed immediately with acute myocardial infarction (AMI) and will be to transported as fast as possible to the coronary care unit. The blood samples retrieved in the ambulance are transported to the lab and to the table top radiometer in the emergency unit. As stated before, an increasing number of patients with AMI are presenting without significant abnormalities on ECG. Therefore, the troponin-T levels in the blood sample will provide extra information to make an appropriate diagnosis. It is our hypothesis, that the Cobas h232 device will provide faster results and thus a faster diagnosis of AMI which benefit patients' outcome.

ELIGIBILITY:
Inclusion Criteria:

* Non-traumatic thoracic pain
* Transportation via ambulance or MUG
* Written informed consent form (ICF) has to be obtained from the patient

Exclusion Criteria:

* Age <18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
The time to diagnosis of acute myocardial infarction (AMI) | one hour
  The time between blood sample and the result of each device will be compared against the other devices. According to the troponin level, the diagnosis will be made. Troponin T< 5 ng/L: negative for AMI; Troponin-T>50 ng/L: positive for AMI; Troponin-T: 5-50 ng/L: observation and a second blood sample has to be taken for re-evaluation of troponin-T.

SECONDARY OUTCOMES:
Time since onset of chest pain to first blood sample | one hour
  The time since onset of chest pain will be asked to the patient. The faster a patient will call to the emergency unit, the better the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Vanelderen, MD PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium